CLINICAL TRIAL: NCT01451060
Title: Maternal and Neonatal Outcomes After the Use of Vasopressors to Correct Hypotension During Cesarean Section Under Spinal Anesthesia in Pregnant Women With Severe Preeclampsia: Randomized Clinical Trial
Brief Title: Maternal and Neonatal Outcomes of the Use of Vasopressors to Treat Hypotension During Spinal Anesthesia for Cesarean
Acronym: Vasopressors
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: We didn't have enough financial support
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Flavia orange, Principal Investigator, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2300-11
Record Dates: First submitted 2011-08-01; First posted 2011-10-13 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2011-10

CONDITIONS: Preeclampsia; Pregnancy Toxemias
Keywords: vasopressors; cesarean anesthesia; hypotension
MeSH Terms: conditions — Pre-Eclampsia; Hypotension | interventions — Metaraminol; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Metaraminol — It will be used a dose of 0.5 mg to any fall in blood pressure of the fetus until birth
  Other Names: Aramin
Drug: Ephedrine — It will be used at any one dose de1mg fall in blood pressure of the fetus until birth
  Other Names: Ephedrin

SUMMARY:
Anesthesia for cesarean section has been a great challenge for the anesthesiologist, for mother and fetus are closely related. So the challenge is to anesthetize the mother without interfering with the physiology of the fetus. The spinal block, although safe, are not free of complications if not treated properly, may be responsible for increased fetal morbidity. Among the major side effects, there is hypotension, with potentially serious consequences for the maternal-fetal dyad. Hypotension in pregnant women at low risk may not lead to major damage, but a pregnant woman with low reserves, as is the case of pregnant women with pre-eclampsia, any drop in blood pressure of the mother can bring harm to the welfare of mother and fetus. Based on the above, the purpose of this study is to compare the effects of maternal and perinatal treatment of hypotension with ephedrine or metaraminol in pregnant women with severe preeclampsia undergoing cesarean section under spinal anesthesia. There will be a randomized, double-blind, which will be included pregnant women with severe preeclampsia with indication of cesarean section, gestational age above 34 weeks gestation and only.Will be Excluded women with hemorrhagic syndromes of pregnancy, HELLP syndrome, eclampsia, cardiovascular or cerebrovascular disease, fetal distress and absolute contraindications to spinal anesthesia.

All patients are fully informed of the research objectives and will only be included in the study if they agree to participate and sign the Instrument of Consent. The project was designed following the recommendations of Resolution 196/96 of the National Health and the Declaration of Helsinki for research involving human subjects (2000). In addition, the project was submitted to the Ethics Committee in Research of the Institute of Integrative Medicine Professor Fernando Figueira, is approved. The study will be conducted from June 2011 to July 2012. The study variables are: consumption of metaraminol and ephedrine before and after birth, the occurrence of nausea and vomiting, incidence of maternal hypotension, the occurrence of reactive hypertension, occurrence of bradycardia, pH of umbilical cord, Apgar score 5 minutes, need for face mask ventilation and ICU admission.

DETAILED DESCRIPTION:
Ephedrine, a long time was considered the safest drug for both mother and fetus during the treatment of hypotension in Caesarean section. However, recent evidence shows that contrary to what was thought, ephedrine appears to increase fetal metabolism, decreasing the pH and excess base.

Recently, phenylephrine has been used in the treatment of hypotension during cesarean delivery with better results in relation to acid-base parameters in umbilical cord blood. However, few data are available on the use of phenylephrine in high-risk pregnancy, the majority of studies in healthy pregnant women for elective caesarean section.

Although little scientific evidence regarding the use of metaraminol for treatment of hypotension in Caesarean section, recent study demonstrated superiority of this drug compared to ephedrine, checking a lower incidence of neonatal acidosis and better control of blood pressure. The researchers also found differences in blood gases from the umbilical cord between the ephedrine and metaraminol groups larger than those already found in previous studies comparing ephedrine and phenylephrine.

The pathophysiological changes in patients with pre-eclampsia can lead to intrauterine growth restriction with chronic fetal distress, due to the limited uteroplacental flow, which, in certain situations, may be reduced by 50% to 70%. Added to this, spinal anesthesia may cause sudden hypotension and fetal acidosis more often, even in elective operations, compared to epidural or general anesthesia, and that these changes may not have clinical significance in healthy fetuses at term, but may be critical in situations where arterial insufficiency uteroplacental and fetal distress already to present. It is believed, therefore, important that treat or prevent hypotension in patients with severe preeclampsia under spinal anesthesia.

Prevention of hypotension in patients with severe preeclampsia does not require large amounts of intravenous fluids, but careful prophylaxis of postural hypotensive syndrome. Despite the care, if hypotension occurs, aggressive treatment is mandatory in these patients and fast in order to avoid worsening fetal distress and neonatal depression. Such patients are more sensitive to vasopressors, therefore, small doses should be administered.

However, the biggest challenge of the anesthesiologist is to determine the ideal vasopressor in pregnant women at high risk, able to adequately restore blood pressure levels without determining deterioration of fetal status.

30 Reynolds and Seed in 2005 showed that ephedrine, administered in large doses, has contributed to the adverse effects of spinal anesthesia (greater degree of fetal metabolic acidosis), supporting the idea that ephedrine is not the vasopressor of choice for treatment of maternal hypotension during cesarean section.

As a result, this study is to fill this knowledge gap, taking on great importance to evaluate maternal and perinatal outcomes of pregnant women with severe preeclampsia to receive ephedrine or metaraminol for treatment of maternal hypotension during caesarean section under spinal anesthesia. Considering the importance of creating a protocol, since the metaraminol, unlike phenylephrine, is widely available at our facility.

ELIGIBILITY:
Inclusion Criteria:

* Severe preeclampsia with indication of cesarean section
* Informed consent for study participation
* Age above 34 weeks gestational
* Single Pregnancy

Exclusion Criteria:

* Hemorrhagic syndromes of pregnancy (placenta previa, DPPNI)
* Help Syndrome
* Eclampsia
* Cardiovascular or Cerebrovascular Disease
* Fetal distress Absolute contraindications to spinal anesthesia (coagulopathy, sepsis and hypovolemia)
* Pregnant unable to decide on participation in the study (unconscious, confused, coma, mental retardation)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of maternal hypotension | During the caesarean, on average during the first 30 minutes after spinal anesthesia
  Participants are accompanied throughout their cesarean section an average of 30 minutes, where they will be measured blood pressure and heart rate every three minutes until the end of cesarean section.

SECONDARY OUTCOMES:
Maternal and Neonatal outcomes | During the cesarean section and postpartum until discharge (an average of 24 hours)
  After the birth of neonatal up to the high infant, an average of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Monteiro, MD, Study Director — Instituto de Medicina integral Professor Fernando Figueira
Locations (1):
- Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We don't have data to share